CLINICAL TRIAL: NCT05566392
Title: Longterm Influence of Pediatric Long COVID Syndrome on the Neuropsychiatric Function, Social Function, Neuroimage, and Gut Microbiota
Brief Title: Longterm Influence of Pediatric Long COVID Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202208086RIND
Record Dates: First submitted 2022-10-02; First posted 2022-10-04 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: COVID-19-Associated Encephalitis; Long COVID
Keywords: pediatric neurology; psychiatric evaluation; Long COVID syndrome; magnetic resonance image
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronavirus disease (COVID): Pediatric patients who was diagnosed as COVID
  Interventions: Diagnostic Test: Brain MRI
- Healthy: Pediatric participants who hadn't been diagnosed COVID before
  Interventions: Diagnostic Test: Brain MRI

INTERVENTIONS:
Diagnostic Test: Brain MRI — Brain MRI including diffusion spectrum image, and functional MRI Interview with questionnaires for neuropsychiatric evaluation Near infrared spectroscopy and resting-state connectivity evaluation
  Other Names: Neuropsychiatric evaluation; Near infrared spectroscopy

SUMMARY:
We enroll pediatric patients who were diagnosed COVID-19 for main observation target. We will perform brain MRI and neuropsychiatric evaluation 4-6 months after COVID-19 diagnosed. We also enroll healthy age- and gender-matched participant for cross-over comparison. We will perform same evaluation process one year later for longitudinal evaluation

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years old
* Has been diagnosed COVID-19 before

Exclusion Criteria:

* History of neuropsychiatric disorders
* Have some device not allowed for MRI

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Aged between 6-18 years old pediatric patient diagnosed as COVID would be enrolled. The patient who had neuropsychiatric disorders would be excluded. We also enroll age- and gender-matched healthy participants for cross-over comparison
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Difference between COVID and healthy group | 1 years after enrollment for primary evaluation
  The neuroimage difference between COVID and healthy group and the correlation with neuropsychiatric evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Tso Lee, PHD, Principal Investigator — National Taiwan University Children Hospital Pediatric neurology department
Locations (1):
- National Taiwan University Children Hospital Pediatric Neurology Department, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
according to our participant consent, the participant information will be stored as de-identification data